CLINICAL TRIAL: NCT00820079
Title: A Phase 2B, Randomised, Double-blind, Placebo-controlled, Parallel Group, Multi-centre Study to Investigate the Efficacy, Mechanism of Action, Pharmacokinetics, Safety and Tolerability of the mGluR5 Negative Allosteric Modulator ADX10059 as Monotherapy in Patients With Gastroesophageal Reflux Disease (GERD)
Brief Title: ADX10059 as a Monotherapy in Patients With Gastroesophageal Reflux (GERD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Addex Pharma S.A. (Industry)
Responsible Party: Study Director, Addex Pharma SA
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADX10059-204; 2008-005104-10
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-12

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastroesophageal reflux; Heartburn; Regurgitation
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADX10059 120 mg (Experimental): Twice-daily
  Interventions: Drug: ADX10059
- ADX10059 Matching Placebo (Placebo Comparator): twice-daily
  Interventions: Drug: ADX10059 Matching Placebo

INTERVENTIONS:
Drug: ADX10059 — oral administration
  Arms: ADX10059 120 mg
Drug: ADX10059 Matching Placebo — oral administration
  Arms: ADX10059 Matching Placebo

SUMMARY:
Evaluation of the effect of ADX10059 on symptom control in patients with gastroesophageal reflux.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of typical GERD
* well controlled on a standard clinical symptoms controlled dose of PPI treatment
* body mass index ≤32 kg/m2

Exclusion Criteria:

* exclusively atypical symptoms of GERD
* symptoms that have been shown not to be associated with GERD
* erosive oesophagitis
* hiatus hernia > 3 cm
* current diagnosis of co-existing psychiatric disease
* known clinically significant allergy or known hypersensitivity to drugs
* pregnant or breast-feeding
* has received sodium valproate or topiramate within 30 days of Screening
* has a history of a significant medical condition that may affect the safety of the patient or preclude adequate participation in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Number of GERD symptom free days in week 2 of study medication treatment | 2 weeks

SECONDARY OUTCOMES:
GERD symptoms | 2 weeks
Sleep disturbance | 2 weeks
Use of antacid rescue medication | 2 weeks
Global assessment of GERD | 2 weeks
Effect on lower oesophageal sphincter and reflux episodes | 2 weeks

CONTACTS AND LOCATIONS:
Locations (11):
- Wien, Vienna, Austria
- Leuven, Leuven, Belgium
- France (3):
  - Bordeaux, Bordeaux
  - Lyon, Lyon
  - Nantes, Nantes
- Germany (6):
  - Berlin, Berlin
  - Dresden, Dresden
  - Gorlitz, Görlitz
  - Leipzig, Leipzig
  - Madgeburg 12, Magdeburg
  - Magdeburg 13, Magdeburg

REFERENCES:
- [Derived] Zerbib F, Bruley des Varannes S, Roman S, Tutuian R, Galmiche JP, Mion F, Tack J, Malfertheiner P, Keywood C. Randomised clinical trial: effects of monotherapy with ADX10059, a mGluR5 inhibitor, on symptoms and reflux events in patients with gastro-oesophageal reflux disease. Aliment Pharmacol Ther. 2011 Apr;33(8):911-21. doi: 10.1111/j.1365-2036.2011.04596.x. Epub 2011 Feb 14. PMID 21320138